CLINICAL TRIAL: NCT02373527
Title: Strict Versus No Fasting Prior to Cardiac Catheterization: A Prospective Evaluation of Safety and Clinical Outcomes
Brief Title: Can we Safely Have Our Patients Eat With Cardiac Catheterization - Nix Or alloW: The CHOW NOW Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Guthrie Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1411-60
Record Dates: First submitted 2015-02-23; First posted 2015-02-27 (Estimated); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Chest Pain
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard - Strict Fasting (No Intervention): No food after midnight the night before the procedure and will be allowed to drink clear liquids up to 2 hours prior to the procedure.
- Non Fasting (Experimental): No Fasting prior to catheterization. Usual meal on the day of the procedure and allowed to drink as usual.
  Interventions: Other: No Fasting prior to catheterization

INTERVENTIONS:
Other: No Fasting prior to catheterization — No restriction for oral intake
  Arms: Non Fasting

SUMMARY:
The purpose of this study is to compare the safety and effects of fasting or not fasting overnight before a cardiac catheterization (heart procedure). The study will compare patients who have nothing to eat after midnight before the procedure to those who are allowed to eat or drink before the procedure.

DETAILED DESCRIPTION:
For years it has been common to have patients fast before a cardiac catheterization. It is believed that fasting may lower the risks of upset stomach, vomiting, and aspiration (stomach contents going to the lungs). New findings show that fasting before the procedure may not be needed. This study will look at the safety and possible benefits of not fasting.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are planned for coronary angiogram or percutaneous intervention, either as outpatients or inpatients

Exclusion Criteria:

* Subjects undergoing emergent procedures or requiring post procedure emergent cardiothoracic surgery
* Pregnant Women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 619 (Actual)
Dates: Start 2015-03-18 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-06-05 (Actual)

PRIMARY OUTCOMES:
Composite incidence of contrast induced nephropathy, peri procedural hypotension, aspiration pneumonia/pneumonitis, nausea, vomiting, hyperglycemia and hypoglycemia | 72 hours

SECONDARY OUTCOMES:
Patient Satisfaction score | 72 hours
Total cost of hospitalization | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Sporn, MD, Principal Investigator — The Guthrie Clinic; Abhishek Mishra, MD, Principal Investigator — The Guthrie Clinic
Locations (1):
- Robert Packer Hospital, Sayre, Pennsylvania, United States